CLINICAL TRIAL: NCT05332080
Title: FUNCTIONAL RECOVERY AFTER A TELEREHABILITATION PROGRAM IN PATIENTS WITH DISTAL RADIUS FRACTURE: A RANDOMIZED CLINICAL TRIAL
Brief Title: Telerehabilitation in Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Juan Figueroa-García, Principal investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2020-3201-153
Record Dates: First submitted 2022-04-05; First posted 2022-04-18 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Distal Radius Fracture
Keywords: Telerehabilitation; physical therapy; distal radius fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, parallel-treatment trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation via application on cell phone (Experimental): The patients in this group had application installed on their cell phones to access the online content, where they received advice on self-care and the type of exercises to be performed. The program consisted of hydrotherapy, mobility exercises, muscle strengthening, and activities to improve wrist and hand function, with planned 4-week objectives. Participants in both groups were provided with written exercise material, training, and advice on how to return to work and leisure activities. Each patient made a weekly record of the therapy he/she performed, including the day, type, and time of development of his/her exercises
  Interventions: Procedure: Telerehabilitation via application on cell phone
- In-person rehabilitation (No Intervention): The patients in this group received an in-person rehabilitation program and was considered the control group, this group received for two weeks a 10-session program for two weeks that included external heat application, stretching, mobilization, strengthening, and occupational therapy. Moreover, it was complemented with occupational therapy focused on improving essential functions and strengthening extrinsic and intrinsic hand musculature, effectiveness in wrist mobility, and simulation of specific activities for reincorporation to work

INTERVENTIONS:
Procedure: Telerehabilitation via application on cell phone — Realization of rehabilitation through content in an app they received advice on self-care and the type of exercises to do. The program consisted of hydrotherapy, mobility exercises, muscle strengthening, and activities to improve wrist and hand function, with planned goals.
  Arms: Telerehabilitation via application on cell phone

SUMMARY:
Objective: To determine the effectiveness of telerehabilitation versus supervised therapy in the functional recovery of patients with distal radius fracture.

Design: A randomized, controlled, parallel-treatment trial protocol was performed to compare functional recovery after a telerehabilitation program vs supervised rehabilitation in patients with distal radius fracture.

Setting:

Participants: A total of 91 patients with distal radius fractures grades AO23 A and B.

Interventions: the supervised rehabilitation group received for two weeks a 10-session program that included external heat application, stretching, mobilization, strengthening, and occupational therapy. The telerehabilitation group was given instructions to apply hydrotherapy, perform mobility and wrist and hand strengthening exercises for four weeks, using the Moodle application on their cell phone.

Main outcomes measures: Outcome measures were measured at the time of admission to rehabilitation and 1, 3, and 6 months; at each follow-up visit, functionality, active range of motion, fist grip strength, quality of life and pain were measured.

Results: When the results obtained at the beginning and at six months were compared, both groups presented statistically significant changes in the clinical variables analyzed but with greater functionality in the telerehabilitation group.

DETAILED DESCRIPTION:
Distal radius fractures (DRF) are among the most frequent fractures worldwide; in the United States, they are the second most common fracture in the upper limb, present an estimated annual incidence of 643,000 and represent 1.5% of consultations for hand and forearm fractures in emergency departments, after fractures of the radius and ulna. Their care implies an increase in the cost of care. In the United Kingdom, the National Health Services estimated an average expenditure of £1375.34 per day/patient, with surgical fixation of the FDR; in the USA, the Medicare system estimated a cost of more than $170 million for the care of these fractures. These patients are usually routinely referred to rehabilitation services after a variable period of immobilization, which increases the cost of care, with inpatient physiotherapy estimated to cost £82.03 per day and outpatient physiotherapy £40.70.

Despite various studies, it is still unclear which type of therapy has the most significant impact on the recovery of wrist function, range of motion, and strength. Currently, studies are showing that home programs are as effective as supervised rehabilitation programs; however, other studies show the opposite.

The Coronavirus disease (COVID-19) pandemic has imposed new paradigms of care for FDR, and now it is recommended to treat it as non-urgent and conservatively. Hence, it is necessary to establish rehabilitation strategies to continue caring for patients without exposing them to the risk of infection. In this sense, the World Confederation of Physical Therapy has proposed the digital practice of rehabilitation services (telemedicine). Therefore, the objective of this study was to determine the effectiveness of telerehabilitation versus supervised therapy in the functional recovery of patients with distal radius fractures.

Material and methods:

Approval was obtained for this study from the institutional review boards of the Hospital General Regional No.1 (R-2020-3201-153) and all patients consented to participate in the study and publication of the results.

Study Design and Intervention:

A randomized, controlled, parallel-treatment trial protocol was performed by using a computer-generated random number of table and concealed allocation (sequential, sealed envelopes filled by a person unconnected with the study), administered by the project coordinator after subject enrollment. Due to the nature of the intervention, neither the subjects nor the investigators were blinded to the intervention.

The first group received an in-person rehabilitation program and was considered the control group, this group received for two weeks a 10-session program for two weeks that included external heat application, stretching, mobilization, strengthening, and occupational therapy. Moreover, it was complemented with occupational therapy focused on improving essential functions and strengthening extrinsic and intrinsic hand musculature, effectiveness in wrist mobility, and simulation of specific activities for reincorporation to work.

The second group members had the Moodle application installed on their cell phones to access the online content, where they received advice on self-care and the type of exercises to be performed. The program consisted of hydrotherapy, mobility exercises, muscle strengthening, and activities to improve wrist and hand function, with planned 4-week objectives. Participants in both groups were provided with written exercise material, training, and advice on how to return to work and leisure activities. Each patient made a weekly record of the therapy he/she performed, including the day, type, and time of development of his/her exercises.

Patient Sample and Setting:

During the period November 2020 - April 2021, men and women older than 15 years were included, with closed distal radius fracture type AO23 A and B, after immobilization for six weeks (with or without surgical fixation), with indication by the orthopedic physician to perform rehabilitation, and who had a cell phone and internet access. Patients with distal radius fractures were excluded if they had any of the following radiographic findings: volar tilt >12°, radial tilt >23° and radial height >12 mm, patients with neurological problems, illiteracy, presence of pressure ulcers in the distal third of the forearm or hand that did not heal, users of orally or intravenously administered steroids, patients with pre-existing and concomitant arthritis or osteoarthritis of the wrist, or history of injury. Subjects with less than 80% adherence to treatment were eliminated.

Sample size calculation:

Fourteen points minimum difference on the Disabilities of the Arm, Shoulder, and Hand (DASH) scale, standard deviation of 20, a significance level of 5%, power of 80%, and an estimated loss of 20% were considered for the sample size calculation. The sample size was 44 subjects per group.

Procedures and equipment:

Each patient was assigned a folio number, integrating his or her file with sociodemographic, clinical, and functional data, obtained through the DASH, quality of life was measured with the 36-Item Short Form Survey (SF-36), for the measurement of the range of movement of the wrist, a commercial goniometer was used, and for the measurement of, the CAMRY electronic hand dynamometer, model: EH101 was used; for everyone, the arithmetic mean was calculated after three consecutive attempts, maintaining the maximum grip strength for 4 seconds, with an interval of 1 minute, as previously described, and for the evaluation of pain, the visual analog scale (VAS) was used.

Outcome assessment:

All participants were assessed for function, range of movement of the wrist, FPP, quality of life and pain at baseline and subsequently at 4, 12, and 24 weeks, irrespective of the degree of compliance with the experimental protocols.

Adherence: All the patients in group 1 reported having attended their therapies on time in their registry card, concluding the treatment cycles. In group 2, adherence was estimated to be between 80-90%, as evidenced by the number of clicks, the number of reproductions of each video, and the average time spent on the portal. The patients had to repeat the exercises at home daily, monitored with telephone calls, exercise diary, and checklist.

Statistical analysis:

Qualitative variables were analyzed with absolute and relative frequencies, quantitative variables with measures of central tendency and dispersion; for the comparison of quantitative variables between groups at the end of treatment, Student's t was used for independent samples.

The student T-test for paired samples was used to analyze intragroup dependent variables at the beginning and end of follow-up. Statistical significance was established at p<0.05. IBM-SPSS Software® v21 statistical/computer program was used for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 15 years
* With closed distal radius fracture type AO23 A and B
* Immobilization for six weeks (with or without surgical fixation)
* With indication by the orthopedic physician to perform rehabilitation
* Have a cell phone and internet access

Exclusion Criteria:

* Patients with distal radius fractures with any of the following radiographic findings: volar tilt >12°, radial tilt >23° and radial height >12 mm
* Patients with neurological problems, illiteracy, presence of pressure ulcers in the distal third of the forearm or hand that did not heal, users of orally or intravenously administered steroids, patients with pre-existing and concomitant arthritis or osteoarthritis of the wrist, or history of injury. Subjects with less than 80% adherence to treatment were eliminated.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Outcome of baseline measures of wrist function and changes at 4, 12 and 24 weeks | At baseline and subsequently at 4, 12, and 24 weeks
  The measures physical function and symptoms in people with musculoskeletal disorders of the upper limb, specifically the wrist, was measured with Disabilities of the Arm, Shoulder and Hand questionnaire, a higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability. The score test ranges from 0 (no disability) to 100 (most severe disability)

SECONDARY OUTCOMES:
Outcome of baseline measures of quality of life and changes at 4, 12 and 24 weeks | At baseline and subsequently at 4, 12, and 24 weeks
  Quality of life is an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. It is a broad ranging concept affected in a complex way by the person's physical health, psychological state, personal beliefs, social relationships and their relationship to salient features of their environment. The 36-item Short Form Survey was used for measure quality of life, with a test score ranging from 0 (worst quality of life) to 100 (best quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano del Seguro Social, HGR 1, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mauck BM, Swigler CW. Evidence-Based Review of Distal Radius Fractures. Orthop Clin North Am. 2018 Apr;49(2):211-222. doi: 10.1016/j.ocl.2017.12.001. PMID 29499822
- [Background] Chung KC, Spilson SV. The frequency and epidemiology of hand and forearm fractures in the United States. J Hand Surg Am. 2001 Sep;26(5):908-15. doi: 10.1053/jhsu.2001.26322. PMID 11561245
- [Background] Tubeuf S, Yu G, Achten J, Parsons NR, Rangan A, Lamb SE, Costa ML. Cost effectiveness of treatment with percutaneous Kirschner wires versus volar locking plate for adult patients with a dorsally displaced fracture of the distal radius: analysis from the DRAFFT trial. Bone Joint J. 2015 Aug;97-B(8):1082-9. doi: 10.1302/0301-620X.97B8.35234. PMID 26224825
- [Background] Shauver MJ, Yin H, Banerjee M, Chung KC. Current and future national costs to medicare for the treatment of distal radius fracture in the elderly. J Hand Surg Am. 2011 Aug;36(8):1282-7. doi: 10.1016/j.jhsa.2011.05.017. Epub 2011 Jun 25. PMID 21705154
- [Background] Wong JY. Time off work in hand injury patients. J Hand Surg Am. 2008 May-Jun;33(5):718-25. doi: 10.1016/j.jhsa.2008.01.015. PMID 18590855
- [Background] Krischak GD, Krasteva A, Schneider F, Gulkin D, Gebhard F, Kramer M. Physiotherapy after volar plating of wrist fractures is effective using a home exercise program. Arch Phys Med Rehabil. 2009 Apr;90(4):537-44. doi: 10.1016/j.apmr.2008.09.575. PMID 19345766
- [Background] Maciel JS, Taylor NF, McIlveen C. A randomised clinical trial of activity-focussed physiotherapy on patients with distal radius fractures. Arch Orthop Trauma Surg. 2005 Oct;125(8):515-20. doi: 10.1007/s00402-005-0037-x. Epub 2005 Oct 22. PMID 16136342
- [Background] Oskarsson GV, Hjall A, Aaser P. Physiotherapy: an overestimated factor in after-treatment of fractures in the distal radius? Arch Orthop Trauma Surg. 1997;116(6-7):373-5. doi: 10.1007/BF00433993. PMID 9266044
- [Background] Watt CF, Taylor NF, Baskus K. Do Colles' fracture patients benefit from routine referral to physiotherapy following cast removal? Arch Orthop Trauma Surg. 2000;120(7-8):413-5. doi: 10.1007/pl00013772. PMID 10968529
- [Background] Handoll HH, Elliott J. Rehabilitation for distal radial fractures in adults. Cochrane Database Syst Rev. 2015 Sep 25;2015(9):CD003324. doi: 10.1002/14651858.CD003324.pub3. PMID 26403335
- [Background] Tenforde AS, Iaccarino MA, Borgstrom H, Hefner JE, Silver J, Ahmed M, Babu AN, Blauwet CA, Elson L, Eng C, Kotler D, Homer S, Makovitch S, McInnis KC, Vora A, Borg-Stein J. Telemedicine During COVID-19 for Outpatient Sports and Musculoskeletal Medicine Physicians. PM R. 2020 Sep;12(9):926-932. doi: 10.1002/pmrj.12422. Epub 2020 Jul 10. PMID 32424977
- [Background] Turolla A, Rossettini G, Viceconti A, Palese A, Geri T. Musculoskeletal Physical Therapy During the COVID-19 Pandemic: Is Telerehabilitation the Answer? Phys Ther. 2020 Aug 12;100(8):1260-1264. doi: 10.1093/ptj/pzaa093. No abstract available. PMID 32386218
- [Background] Gunther CM, Burger A, Rickert M, Crispin A, Schulz CU. Grip strength in healthy caucasian adults: reference values. J Hand Surg Am. 2008 Apr;33(4):558-65. doi: 10.1016/j.jhsa.2008.01.008. PMID 18406961
- [Background] Egund L, Onnby K, Mcguigan F, Akesson K. Disability and Pain are the Best Predictors of Sick Leave After a Distal Radius Fracture in Men. J Occup Rehabil. 2020 Dec;30(4):656-664. doi: 10.1007/s10926-020-09880-4. PMID 32052265
- [Background] Azad A, Kang HP, Alluri RK, Vakhshori V, Kay HF, Ghiassi A. Epidemiological and Treatment Trends of Distal Radius Fractures across Multiple Age Groups. J Wrist Surg. 2019 Aug;8(4):305-311. doi: 10.1055/s-0039-1685205. Epub 2019 Apr 16. PMID 31404224
- [Background] Rundgren J, Bojan A, Mellstrand Navarro C, Enocson A. Epidemiology, classification, treatment and mortality of distal radius fractures in adults: an observational study of 23,394 fractures from the national Swedish fracture register. BMC Musculoskelet Disord. 2020 Feb 8;21(1):88. doi: 10.1186/s12891-020-3097-8. PMID 32035488
- [Background] Sander AL, Leiblein M, Sommer K, Marzi I, Schneidmuller D, Frank J. Epidemiology and treatment of distal radius fractures: current concept based on fracture severity and not on age. Eur J Trauma Emerg Surg. 2020 Jun;46(3):585-590. doi: 10.1007/s00068-018-1023-7. Epub 2018 Oct 1. PMID 30276724
- [Background] Wakefield AE, McQueen MM. The role of physiotherapy and clinical predictors of outcome after fracture of the distal radius. J Bone Joint Surg Br. 2000 Sep;82(7):972-6. doi: 10.1302/0301-620x.82b7.10377. PMID 11041584
- [Background] Challis MJ, Jull GJ, Stanton WR, Welsh MK. Cyclic pneumatic soft-tissue compression enhances recovery following fracture of the distal radius: a randomised controlled trial. Aust J Physiother. 2007;53(4):247-52. doi: 10.1016/s0004-9514(07)70005-3. PMID 18047459
- [Background] Kay S, Haensel N, Stiller K. The effect of passive mobilisation following fractures involving the distal radius: a randomised study. Aust J Physiother. 2000;46(2):93-101. doi: 10.1016/s0004-9514(14)60317-2. PMID 11676793
- [Background] Lara TR, Kagan RP, Hiratzka SL, Thompson AR, Nazir OF, Mirarchi AJ. Traditional Versus Digital Media-Based Hand Therapy After Distal Radius Fracture. J Hand Surg Am. 2022 Mar;47(3):291.e1-291.e8. doi: 10.1016/j.jhsa.2021.06.018. Epub 2021 Aug 6. PMID 34366180
- [Background] Andrade-Silva FB, Rocha JP, Carvalho A, Kojima KE, Silva JS. Influence of postoperative immobilization on pain control of patients with distal radius fracture treated with volar locked plating: A prospective, randomized clinical trial. Injury. 2019 Feb;50(2):386-391. doi: 10.1016/j.injury.2018.12.001. Epub 2018 Dec 4. PMID 30558805
- [Background] Pasila M, Sundholm A. Mobilization of stiff hands after 104 Colles' fractures: a comparison between the value of the Movelat and its base cream. Rheumatol Rehabil. 1980 Aug;19(3):170-2. doi: 10.1093/rheumatology/19.3.170. No abstract available. PMID 7414186
- [Background] Lyngcoln A, Taylor N, Pizzari T, Baskus K. The relationship between adherence to hand therapy and short-term outcome after distal radius fracture. J Hand Ther. 2005 Jan-Mar;18(1):2-8; quiz 9. doi: 10.1197/j.jht.2004.10.008. PMID 15674780
- [Background] Souer JS, Buijze G, Ring D. A prospective randomized controlled trial comparing occupational therapy with independent exercises after volar plate fixation of a fracture of the distal part of the radius. J Bone Joint Surg Am. 2011 Oct 5;93(19):1761-6. doi: 10.2106/JBJS.J.01452. PMID 22005860
- [Background] Upadhyaya GK, Iyengar K, Jain VK, Vaishya R. Challenges and strategies in management of osteoporosis and fragility fracture care during COVID-19 pandemic. J Orthop. 2020 Jun 2;21:287-290. doi: 10.1016/j.jor.2020.06.001. eCollection 2020 Sep-Oct. PMID 32523258
- [Background] Moore CM, Leonardi-Bee J. The prevalence of pain and disability one year post fracture of the distal radius in a UK population: a cross sectional survey. BMC Musculoskelet Disord. 2008 Sep 29;9:129. doi: 10.1186/1471-2474-9-129. PMID 18823546
- [Background] MacIntyre NJ, Dewan N. Epidemiology of distal radius fractures and factors predicting risk and prognosis. J Hand Ther. 2016 Apr-Jun;29(2):136-45. doi: 10.1016/j.jht.2016.03.003. PMID 27264899